CLINICAL TRIAL: NCT00787241
Title: Platelet Count Trends in Pre-eclamptic Parturients: What is the Predictive Value of an Initial Platelet Count During Labor?
Brief Title: Platelet Count Trends in Pre-eclamptic Parturients
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Cynthia Wong, Professor of Anesthesiology, Northwestern University
Other Study IDs: 0524-015
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Results first posted 2012-02-17 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Obstetric Labor Complications; Preeclampsia; Thrombocytopenia
Keywords: Platelets; Labor; Preeclampsia
MeSH Terms: conditions — Obstetric Labor Complications; Pre-Eclampsia; Thrombocytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Mild preeclampsia: Preeclampsia without eclampsia or HELLP syndrome
- Severe preeclampsia: Severe preeclampsia with eclampsia and/or HELLP syndrome
- Mild preeclampsia superimposed on chronic hypertension: Mild preeclampsia in association with chronic hypertension

SUMMARY:
Thrombocytopenia (platelet count < 100,000/mL) occurs in approximately 15% of women with preeclampsia. Neuraxial analgesia is contraindicated in parturients with a coagulopathy; therefore, the platelet count(PC) is routinely checked prior to the initiation of neuraxial analgesia in women with preeclampsia/eclampsia. Catheter removal is also contraindicated in the presence of a coagulopathy. Some women have an acceptable PC at the initiation of neuraxial analgesia, but may become significantly more thrombocytopenic during labor and delivery. In a study of severely preeclamptic parturients, some with HELLP (H=hemolysis of red blood cells, EL=elevated liver enzymes, LP=low platelet count) syndrome, the admission PC correlated with the PC nadir. However, the natural progression of the PC has not been studied in women with mild preeclampsia. We hypothesize that women with mild preeclampsia or severe preeclampsia without HELLP syndrome, and whose admission PC is greater than 150,000/mL, will have a stable PC during the course of labor and delivery and do not require another PC check prior to initiation of neuraxial analgesia or removal of the epidural catheter. The purpose of this study is to determine the positive predictive value of an initial PC greater than 150,000/mL for maintaining a PC greater than 80,000/mL during labor and delivery.

DETAILED DESCRIPTION:
All women who delivered from 1/2000 through 12/2002, with the discharge diagnosis of mild preeclampsia, severe preeclampsia (including HELLP and eclampsia), and preeclampsia superimposed on chronic hypertension were identified through the Perinatal Database. Platelet counts (PC) for each patient, from one month prior to the delivery admission, until hospital discharge, were analyzed. The number of PC determinations per parturient was determined. For each diagnosis, the positive predictive value (PPV) of an initial PC > 150,000/mL for maintaining subsequent PC > 80,000/mL, as well as the PPV of the PC prior to initiation of neuraxial analgesia was calculated. The median time interval from the closest PC determination to initiation of neuraxial analgesia was calculated.

ELIGIBILITY:
Inclusion Criteria:

* All participants who delivered between January 1, 2000 and December 31, 2002, identified as having preeclampsia (without HELLP syndrome) in the Perinatal Database.

Exclusion Criteria:

* Participants not diagnosed with preeclampsia and/or outside the given criteria dates.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant Women
Sampling Method: Non-Probability Sample
Enrollment: 445 (Actual)
Dates: Start 2002-09; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Wong, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Weiner CP. Preeclampsia-eclampsia syndrome and coagulation. Clin Perinatol. 1991 Dec;18(4):713-26. PMID 1837248
- [Background] Leduc L, Wheeler JM, Kirshon B, Mitchell P, Cotton DB. Coagulation profile in severe preeclampsia. Obstet Gynecol. 1992 Jan;79(1):14-8. PMID 1727573

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women who delivered from 1/2000 thru 12/2002 with the discharge diagnosis of mild preeclampsia, severe preeclampsia and preeclampsia superimposed on chronic hypertension were retrospectively evaluated.
Groups:
- Mild Preeclampsia: Subjects with a discharge diagnosis of mild preeclampsia
- Severe Preeclampsia: Subjects with a discharge diagnosis of severe preeclampsia including HELP syndrome
- Mild Preeclampsia Superimposed on Chronic Hypertension: Subjects with a discharge diagnosis of preeclampsia with a history of chronic hypertension prior to pregnancy
Period: Overall Study
Arm/Group | Mild Preeclampsia | Severe Preeclampsia | Mild Preeclampsia Superimposed on Chronic Hypertension
Started | 261 | 143 | 41
Completed | 261 | 143 | 41
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild Preeclampsia | Severe Preeclampsia | Mild Preeclampsia Superimposed on Chronic Hypertension | Total
Number analyzed (Participants) | 261 | 143 | 41 | 445
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 261 | 143 | 41 | 445
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 261 | 143 | 41 | 445
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 261 | 143 | 41 | 445

OUTCOME MEASURES:

1. Primary Outcome: Positive Predictive Value of Earliest Available Platelet Count
Description: The positive predictive value of the earliest available platelet count with the maintenance of a platelet count greater than 80,000 during labor and delivery and removal of the epidural catheter was calculated. The test was considered true if the first platelet count was >150,000 platelets and the subsequent platelet counts remained above 80,000 platelets. The number of subjects with a test equal true was divided by the total number of subjects with a platelet counts >150,000 at the earliest available platelet count multiplied by 100.
Time Frame: 0 to 72 hours following delivery
Measure: Number; unit: percentage of positive platelet counts
Groups:
- Severe Preeclampsia: Subjects with a diagnosis of severe preeclampsia at discharge
- Mild Preeclampsia Superimposed on Chronic Hypertension: Subjects with a diagnosis of mild preeclampsia at discharge with a history of chronic hypertension
Arm/Group | Mild Preeclampsia | Severe Preeclampsia | Mild Preeclampsia Superimposed on Chronic Hypertension
Number analyzed (Participants) | 261 | 143 | 41
percentage of positive platelet counts | 99 | 90 | 100

2. Secondary Outcome: Positive Predictive Value of Platelet Count Closet to Neuraxial Analgesia
Description: The positive predictive value of the platelet count closest to neuraxial analgesia with the maintenance of a platelet count greater than 80,000 during labor and delivery and removal of the epidural catheter was calculated. The test was considered true if the closest platelet count was >150,000 platelets and the subsequent platelet counts remained above 80,000 platelets. The number of subjects with a test equal true was divided by the total number of subjects with a platelet counts >150,000 at the closest available platelet count multiplied by 100.
Time Frame: 0 to 72 hours following delivery
Measure: Number; unit: percentage of positive platelet counts
Arm/Group | Mild Preeclampsia | Severe Preeclampsia | Mild Preeclampsia Superimposed on Chronic Hypertension
Number analyzed (Participants) | 261 | 143 | 41
percentage of positive platelet counts | 99 | 93 | 100

3. Secondary Outcome: Time Interval (Hours) From Closet Platelet Count to Initiation of Neuraxial Analgesia
Description: Time interval in hours from the closest obtained platelet count to the initiation of neuraxial analgesia.
Time Frame: 1 week to time of neuraxial analgesia
Measure: Median (Full Range); unit: Hours
Arm/Group | Mild Preeclampsia | Severe Preeclampsia | Mild Preeclampsia Superimposed on Chronic Hypertension
Number analyzed (Participants) | 261 | 143 | 41
Hours | 4 [0.5 to 474] | 3 [0.1 to 35.3] | 4 [0.5 to 42.8]

ADVERSE EVENTS:
Arm/Group | Mild Preeclampsia | Severe Preeclampsia | Mild Preeclampsia Superimposed on Chronic Hypertension
Serious Adverse Events (participants affected / at risk) | 0/261 | 0/143 | 0/41
Other Adverse Events (participants affected / at risk) | 0/261 | 0/143 | 0/41

LIMITATIONS AND CAVEATS:
Retrospective trial and obtaining platelet counts was not done per protocol so cannot predict the greatest interval that is acceptable to demonstrate platelet counts greater than 150,000 during labor and delivery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No